CLINICAL TRIAL: NCT00947609
Title: Improving the Diagnosis and Management of Latent Tuberculosis in Thai Children
Brief Title: Improving Latent Tuberculosis (TB) Diagnosis in Thai Children
Acronym: TB Px
Status: Completed | Type: Observational
Sponsor: SEARCH Research Foundation (Other)
Collaborators: Columbia University (Other); New York Blood Center (Other); HIV Netherlands Australia Thailand Research Collaboration (Network); Queen Sirikit National Institute of Child Health (Other Government)
Responsible Party: Principal Investigator, Hong Van Tieu, Co-investigator, Columbia University
Other Study IDs: SEARCH TB Px
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Latent Tuberculosis; HIV Infections
Keywords: Latent tuberculosis; HIV; Children; Interferon gamma release assays; Thailand; QuantiFERON TB Gold In-tube; T-Spot.TB
MeSH Terms: conditions — Latent Tuberculosis; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infected and HIV-uninfected children: HIV-infected and HIV uninfected children with recent exposure to adults with active tuberculosis will be referred to the two study sites (HIV-NAT/Chulalongkorn and Queen Sirikit) for eligibility screening and enrollment in the study.

SUMMARY:
The study is a prospective study to improve the diagnosis and management of latent TB in HIV-infected and HIV uninfected children in Thailand. The objectives are to assess the sensitivity and specificity of IGRAs (T-Spot®.TB, a T-cell-based assay, and QuantiFERON®-TB Gold In-tube, a whole blood assay), TST, and a refined symptom-based questionnaire in diagnosing latent TB in 166 HIV-infected and HIV uninfected children in Thailand, and to evaluate the influence of age, nutritional and immune status on children's response to the IGRAs. These children will be screened for TB with a detailed TB contact history, symptom-based questionnaire, physical examination, TST, chest radiograph (and abdominal ultrasound for those with abdominal symptoms), IGRAs, and clinical specimens for acid fast bacilli stain and culture. A diagnostic algorithm will be generated using the combination of test modalities with the highest sensitivity and specificity results.

DETAILED DESCRIPTION:
Study Objectives

* To compare the utility of IGRAs, T-Spot®.TB and QuantiFERON®-TB Gold In-Tube, and TST for screening of latent TB in HIV-infected children
* To compare these different screening modalities in HIV-infected children to HIV uninfected children
* To assess the influence of age, nutritional and immune status, prior BCG and TST status on children's response to IGRAs
* To assess the prognostic value of IGRAs vs. TST in predicting development of active TB in children over 9 months

Research questions:

Primary:

What is the sensitivity and specificity of IGRAs and TST in screening for latent TB in HIV-infected and HIV uninfected children in Thailand?

Secondary:

How do age, nutritional and immune status, prior BCG and PPD status influence children's response to IGRAs? What is the prognostic value of IGRAs vs. TST in predicting development of active TB in children over 9 months?

This is a prospective cohort study conducted at two sites in Bangkok, Thailand: HIV Netherlands Australia Thailand (HIV-NAT) Clinic/Chulalongkorn Hospital and Queen Sirikit National Institute of Child Health.

ELIGIBILITY:
Inclusion Criteria:

1. Have close contact with a person > 15 years of age who had active pulmonary (± extrapulmonary), sputum AFB positive TB (household member or non-household member with contact > 120 hours/month) during the past year
2. Are between the ages of 2 months and 16 years
3. Parents or caregivers provide informed consent to participate
4. Provide child assent for children aged ≥ 7 years

Exclusion Criteria:

1. Child and/or parent/caregiver who refuse study participation
2. Are currently receiving antituberculosis medications for TB disease
3. Have recently been diagnosed with active TB within past 6 months

Ages: 2 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Thai children between the ages of 2 months and 16 years with exposure to active TB adult cases will be referred to the two study sites for eligibility screening.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jintanat Ananworanich, MD, PhD, Principal Investigator — South East Asia Research Collaboration with Hawaii, HIV Netherlands Australia Thailand Research Collaboration, Bangkok, Thailand; Piyarat Suntarattiwong, MD, Principal Investigator — Queen Sirikit National Institute of Child Health, Bangkok, Thailand; Simon Tsiouris, MD, MPH, Principal Investigator — Columbia University
Locations (2):
- Thailand (2):
  - HIV Netherlands Australia Thailand (HIV-NAT) Research Organization, Bangkok
  - Queen Sirikit National Institute of Child Health, Bangkok